CLINICAL TRIAL: NCT03663218
Title: PRE-ProstAtectomy MRI-GuidEd Stereotactic Body RadioTherapy for High-Risk Prostate Cancer Trial (PREPARE SBRT)
Acronym: PREPARE SBRT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1712018849
Record Dates: First submitted 2018-08-30; First posted 2018-09-10 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single Arm (Other): This is a modified dose escalation and de-escalation study with an expansion of 3 or 6 pts to allow the recommended phase II dose (RP2D) be examined in a total of 9 pts. The dose limiting toxicity (DLT) is defined as Grade 3 or higher toxicity related to preoperative radiotherapy according to the Clavien-Dindo Classification. 3 radiation dose levels, 5 Gy, 6 Gy and 6.5Gy are considered. At the start of each dose level, 3 pts will be enrolled and treated for five days. If none of the 3 pts develop the DLT, the testing dose will escalate to the next level. If 1 of the 3 pts develops the DLT, the current dose will be tested in an additional 3 pts. If no additional pts develop the DLT, the dose will escalate.
  Interventions: Radiation: Dose escalation

INTERVENTIONS:
Radiation: Dose escalation — This is a modified dose escalation and de-escalation study with an expansion of 3 or 6 pts to allow the recommended phase II dose (RP2D) be examined in a total of 9 pts. The dose limiting toxicity (DLT) is defined as Grade 3 or higher toxicity related to preoperative radiotherapy according to the Clavien-Dindo Classification. 3 radiation dose levels, 5 Gy, 6 Gy and 6.5Gy are considered. At the start of each dose level, 3 pts will be enrolled and treated for five days. If none of the 3 pts develop the DLT, the testing dose will escalate to the next level. If 1 of the 3 pts develops the DLT, the current dose will be tested in an additional 3 pts. If no additional pts develop the DLT, the dose will escalate.

SUMMARY:
Men with prostate cancer with Gleason Score of 8 or greater or clinical/radiographic evidence of T3 disease will be considered for this trial.

DETAILED DESCRIPTION:
Patients with a diagnosis of high risk prostate cancer with a Gleason score of 8 or greater are eligible for this trial. The study will enroll 20 subjects in 3 years. This is a single arm study and the primary objectives is to assess if a patient can undergo a radical prostatectomy after SBRT without a post-operative grade 3 or higher toxicity (according to Clavien-Dindo Classification) at 30 days. Secondary objectives are to assess acute toxicity and quality of life scores. Exploratory objectives will include analysis of tumor and normal biopsied and resected tissue and serum markers and interpretation of interfraction and intrafraction MRIs.

ELIGIBILITY:
Inclusion Criteria:

* Men aged greater than equal to18 with histologically confirmed primary prostate cancer.
* KPS greater than equal to 70
* Patient with a negative staging bone scan.
* Patient can undergo an MRI.
* Patient with negative staging CT or MRI of pelvis. Suspicious evidence of nodal involvement on staging CT or MRI of pelvis is defined as greater than 1 cm on short axis. Documented negative biopsy of suspicious node required.
* Patient is medically fit to undergo prostatectomy.
* Patient has either Gleason Score greater than equal to 8 on biopsy and/or clinical/radiographic evidence of T3 disease.

Exclusion Criteria:

* Prior history of receiving pelvic radiotherapy.
* Patient is unwilling to undergo prostatectomy.
* Patient with active inflammatory bowel disease defined as currently receiving therapy for IBD.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients with a diagnosis of high risk prostate cancer who meet the inclusion and exclusion criteria will be eligible for participation in this study.
Enrollment: 35 (Estimated)
Dates: Start 2018-10-24 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Number of subjects who successfully complete radical prostatectomy after SBRT without a post-operative DLT of grade 3 or higher | 1 month
  Successful completion of radical prostatectomy after SBRT without a post-operative DLT of grade 3 or higher within 30 days after prostatectomy.

SECONDARY OUTCOMES:
Acute toxicity in patients after stereotactic body radiotherapy (SBRT) and radical prostatectomy (RP) will be assessed based on NCI Common terminology criteria for adverse events (CTCAE) version 5.0. | 3 months
  Acute toxicity in patients after stereotactic body radiotherapy (SBRT) and radical prostatectomy (RP) will be assessed based on NCI Common terminology criteria for adverse events (CTCAE) version 5.0.
Quality of life scores in patients after stereotactic body radiotherapy (SBRT) and radical prostatectomy (RP) will be collected. | 5 years
  Quality of life scores in patients after stereotactic body radiotherapy (SBRT) and radical prostatectomy (RP) will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia C. Formenti, M.D., Principal Investigator — Weill Cornell Medicine - New York Presbyterian Hospital
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No